CLINICAL TRIAL: NCT07103824
Title: Validity and Test-Retest Reliability of Reactive Neurocognitive Upper Extremity Tests in Archers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ebru Tekin, Pamukkale University, Balikesir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024/14
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Athlete Assessment; Archery; Neurocognitive Functional Performance Tests
Keywords: Motor-Cognitive Assessment; Reaction Time; Reactive Upper Limb Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upper Extremity Neurocognitive Tests (Experimental)
  Interventions: Other: Upper Extremity Neurocognitive Tests

INTERVENTIONS:
Other: Upper Extremity Neurocognitive Tests — The validity and test-retest reliability of the Reactive Neurocognitive Upper Extremity Tests (Reactive CKCUEST and Reactive 90/90 Wall Throws Test) will be analyzed through this protocol. Participants will undergo three assessment sessions spaced one week apart: measurements will be conducted using the Catchpad device during the first and third weeks, and the BlazePod™ device during the second week. To ensure blinding, the personnel responsible for conducting the assessments, recording the data, and performing the statistical analyses will be distinct individuals. Participants will be familiarized with the devices one week prior to testing, and a standardized 5-minute free walking warm-up will be administered at each session. All assessments will be performed under similar environmental conditions and at consistent times of day.

SUMMARY:
In archery, the evaluation of reaction time and neurocognitive functions plays a critical role in the management of upper extremity (UE) injuries and return-to-play (RTP) processes. Reaction time reflects an athlete's ability to respond quickly and effectively to visual stimuli, which is particularly crucial in precision-based sports like archery that require high levels of coordination and attention.

With advancements in technology, LED-based systems such as BlazePod™, Catchpad, and ReactionX are increasingly being used in clinical and sports settings to assess cognitive performance and motor responses simultaneously. These tools offer dynamic and motivating methods for evaluating neurocognitive functions. However, before such devices can be reliably used in clinical or research environments, their validity and test-retest reliability must be systematically examined.

The aim of this study is to evaluate the test-retest reliability and validity of Reactive Neurocognitive Upper Extremity Tests-specifically the Reactive Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) and the Reactive 90/90 Wall Throws Test-using the Catchpad system in archers. Based on methodological standards for reliability studies, a minimum of 18 participants will be included. Each participant will attend three test sessions over three weeks: Catchpad in weeks one and three, and BlazePod™ in week two. To ensure blinding, different researchers will conduct the assessments, record the data, and perform the statistical analyses.

Findings from this study are expected to provide scientific evidence supporting the use of Catchpad technology in neurocognitive and reaction time assessments, contributing to more objective decision-making during RTP and potentially reducing the risk of reinjury.

ELIGIBILITY:
Inclusion Criteria:

* Participants must agree to abstain from alcohol and caffeine throughout the study period.
* Participants must refrain from engaging in vigorous physical activity for at least 24 hours prior to each testing session.
* Participants must not consume any food within 3 hours before the measurement.

Exclusion Criteria:

* History of a back, lower extremity, or upper extremity injury within the past six months.
* Any known medical condition or diagnosis that may interfere with testing, including but not limited to neurological disorders.
* Vestibular disorders, color blindness, or the use of medications that could affect balance or visual-motor reaction time.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
REACTIVE CKCUEST+ TEST | three times, one week apart, three-week period
  The test is performed bilaterally twice, each lasting 15 seconds. Three LED lights are arranged with a distance of 36 inches between them. Two LED lights on the same side are positioned 12 inches apart, while a single LED light is placed centrally between the two lights on the opposite side. The LEDs are arranged in a home base pattern, and the lights are configured to change instantaneously upon being touched, with zero delay. The target colors are set as blue for the two LEDs on the same side and red for the single LED on the opposite side. The athlete begins in a high plank position, with hands centered among the LEDs and feet shoulder-width apart. The participant is instructed to stabilize on one arm and sequentially touch the blue LEDs that light up on the same side, followed by the red LED on the opposite side, alternating between the blue and red LEDs using one hand. The objective is to touch as many lights as possible within the allotted time. Upon completion, the total number
REACTIVE 90/90 WALL THROWS TEST | three times, one week apart, three-week period
  This test is performed bilaterally in two trials of 15 seconds each. Three LED lights are vertically aligned on a wall, spaced 12 inches apart. The lights are positioned 6 inches from the corner, with the middle light placed 5 feet above the ground. An identical setup is arranged on the opposite wall or corner for the contralateral limb. The LEDs are programmed so that one target light (blue) illuminates while the other two display random distracting colors. The lights change immediately upon touch with zero delay.
  The athlete stands facing the wall, holding a 2 lb plyoball in 90 degrees of shoulder abduction and 90 degrees of elbow flexion. They are instructed to continuously perform wall throws while maintaining shoulder and elbow alignment, and to touch the target-colored LED as many times as possible with the throwing hand. The non-throwing hand is used to follow the target color. Upon test completion, the total number of touches, number of errors, and average reaction time are r

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University, Balıkesir, Bigadiç, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No